CLINICAL TRIAL: NCT02541643
Title: Expanded Access Single Named Patient Program With Elotuzumab (BMS-901608) for the Treatment of Patient R-A With Relapsed/Refractory Multiple Myeloma
Status: No longer available | Type: Expanded Access
Sponsor: Sundar Jagannath (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Sundar Jagannath, Director of the Multiple Myeloma Program, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Other Study IDs: GCO 14-2022
Record Dates: First submitted 2015-09-02; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Multiple Myeloma
Keywords: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab

INTERVENTIONS:
Drug: Elotuzumab — Elotuzumab will be administered intravenously at a dose of 10mg/kg weekly (Days 1, 8, 15, and 22 of a 4-233k cycle) of the first 2 cycles and every 2 weeks (Day 1 and Day 15) thereafter.
  A window of -1 to +3 days is permitted in Cycles 1 and 2. In Cycle 1 and 2, an elotuzumab dose that falls outside of the pre-specified window must be skipped. In Cycles 3 and beyond, elotuzumab dosing may be delayed for up to 1 week as clinically indicated. If unable to administer within 1 week, then the dose should be skipped and resumption of the elotuzumab continues per the guidance document defined schedule. In addition the following premedication must also be administered 30-90 minutes prior to any elotuzumab:
  * H1 blocker: diphenhydramine (25-50mg PO or IV) or equivalent
  * H2 blocker: ranitidine (50mg IV) or equivalent
  * acetaminophen (650-1000mg PO)
  Other Names: BMS-901608

SUMMARY:
To provide elotuzumab treatment for single-patient use.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent

  a) Before any program procedures are performed, the patient will have the details of the program described to him or her, and she or he will be given a written informed consent document to read. Then, if the patient consents to participate in the program, she or he will indicate that consent by signing and dating the informed consent document in the presence of program personnel.
* Other Criteria

  a) Patients must be willing to refrain from blood donations during program drug therapy and for 8 weeks after therapy.
* Age and Reproductive Status

  1. Men and women, aged 18 years
  2. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
  3. Women must not be breastfeeding
  4. WOCBP must use method(s) of contraception as indicated in the Informed Consent Form. Because of the teratogenic potential of elotuzumab, a highly effective method(s) of contraception (failure rate of less than 1% per year) is required. The individual methods of contraception and duration should be determined in consultation with the investigator. In this study men and WOCBP must be using methods of contraception for at least 1 month (4 weeks) before and women for up to 8 weeks, men for up to 90 days, after the last dose of elotuzumab.
  5. Males who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. The investigator shall review contraception methods and the time period that contraception must be followed. Men that are sexually active with WOCB must agree to follow instructions for method(s) of contraception for the duration of treatment with elotuzumab plus 5 half-lives of the program drug plus 90 days (duration of sperm turnover) for a total of 90 days post-treatment completion.
  6. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile and azoospermic men do not require contraception.

Exclusion Criteria:

* Sex and Reproductive Status

  1. WOCBP not using 2 forms of effective birth control.
  2. Women with a positive pregnancy test at enrollment or prior to administration of program medication.
* Other Exclusion Criteria

  1. Prisoners or patients who are involuntarily incarcerated.
  2. Patients who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Elotuzumab CA204022 BMS-901608 Expanded Access Guidance Document 23 Eligibility criteria for this program have been carefully considered to ensure the safety of the program patients and to ensure that the results of the program can be used. It is imperative that patients fully meet all eligibility criteria.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Sundar Jagannath, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School.of Medicine at Mount Sinai, New York, New York, United States